CLINICAL TRIAL: NCT04374305
Title: Innovative Trial for Understanding the Impact of Targeted Therapies in NF2-Related Schwannomatosis (INTUITT-NF2)
Acronym: INTUITT-NF2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scott R. Plotkin, MD, PhD (Other)
Collaborators: Takeda (Industry); The Children's Tumor Foundation (Other); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor-Investigator, Scott R. Plotkin, MD, PhD, Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-828
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Neurofibromatosis Type 2; Vestibular Schwannoma; Non-vestibular Schwannoma; Meningioma; Ependymoma
Keywords: neurofibromatosis type 2 (NF2); vestibular schwannomas (VS); non-vestibular schwannomas (non-VS); meningioma; ependymoma
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic; Meningioma; Ependymoma | interventions — brigatinib; neratinib

STUDY DESIGN:
Intervention Model Description: The study is a platform-basket trial that includes a Master Protocol with embedded Drug Sub-studies. Currently, there are two drug sub-studies: sub-study A (brigatinib) and sub-study B (neratinib). The overall number of arms is not fixed by design because the investigators include arm-dropping rules for futility and allow for the possibility of arm addition by amendment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sub-study A (brigatinib) - CLOSED TO ENROLLMENT (Experimental): Subjects treated in this arm will receive brigatinib 90 mg by mouth daily for 7 days and then increased to 180 mg by mouth daily if the drug is tolerated.
  Interventions: Drug: Brigatinib
- Sub-study B (neratinib) (Experimental): The first three participants treated in this arm will receive neratinib 200 mg mg by mouth daily. If these participants tolerate the medication well, subsequent participants will receive neratinib 240 mg by mouth daily.
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Brigatinib — Oral daily per predetermined dosage per protocol.
  Other Names: Alunbrig
  Arms: Sub-study A (brigatinib) - CLOSED TO ENROLLMENT
Drug: Neratinib — Oral daily per predetermined dosage per protocol.
  Other Names: Nerlynx
  Arms: Sub-study B (neratinib)

SUMMARY:
This is a multi-arm phase II platform-basket screening study designed to test multiple experimental therapies simultaneously in patients with NF2-related schwannomatosis (NF2-SWN, formerly known as neurofibromatosis type 2) with associated progressive tumors of vestibular schwannomas (VS), non-vestibular schwannomas (non-VS), meningiomas, and ependymomas.

This Master Study is being conducted as a "basket" study that may allow people with multiple tumor types associated with NF2-SWN to receive new drugs throughout this study. Embedded within the Master Study are individual drug substudies.

* Investigational Drug Sub-study A: Brigatinib
* Investigational Drug Sub-study B: Neratinib

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of investigational drugs to learn whether the drug(s) works in treating a specific disease. As a basket study, the trial will enroll patients with NF2-SWN with associated progressive tumors of vestibular schwannomas (VS), non-vestibular schwannomas (non-VS), meningiomas, and ependymomas

The MASTER STUDY is intended to enroll participants who will be allocated into different treatment arms (SUB-STUDIES) which will each have an additional consent and enrollment processes.

MASTER STUDY

-- The research study procedures include screening for eligibility, randomization to an experimental treatment sub-study, if qualified, and observation for up to 10 years.

* Participants who have tumors grow during a treatment sub-study will be permitted to enroll in a different experimental treatment sub-study if they are eligible.
* Participants who are not eligible for enrollment in a different treatment sub-study will be permitted to remain under observation on the Master Study to understand the growth pattern of these tumors (natural history)

  * Participants will be eligible to remain on this Master study for up to 10 years.
  * It is expected that about 80 people will take part in the Master Study
  * The study will randomize a maximum of 40 patients to each of the experimental arms. The overall size of the trial is not fixed by design because it include arm-dropping rules for futility and allow for the possibility of arm addition by amendment.

SUB-STUDY A (brigatinib) Drug Sub-study A will test the activity of brigatinib for treatment of NF2-related tumors.

* Brigatinib is approved for the treatment of people with anaplastic lymphoma kinase (ALK)- positive metastatic non-small cell lung cancer (NSCLC) who have progressed or are intolerant to crizotinib. In preclinical models, brigatinib has shown evidence of activity against models of NF2-deficient tumors.
* Forty (40) people will take part in the Brigatinib Sub-study.
* The sub-study with brigatinib includes two stages.
* In Stage 1, 20 subjects with any allowable tumor type will be accrued to each arm. A minimum of 2 subjects per tumor type (vestibular schwannoma, non-vestibular schwannoma, meningioma, and ependymoma) must be accrued in Stage 1. Interim analysis will be performed after Stage 1 to determine the radiographic response rate (RR) for each tumor types. Subsequently, in stage 2, another 20 subjects will be accrued into the 2 baskets with the most promising early results. If the results are equally promising for more than 2 baskets, subjects will be allocated to the appropriate number of baskets.

SUB-STUDY B (neratinib) Collaborator: National Comprehensive Cancer Network (NCCN) through a grant provided by Puma Biotechnology Drug Sub-study B will test the activity of neratinib for treatment of NF2-related tumors.

* Neratinib is approved for the treatment of people with early stage HER2-overexpressed/amplified breast cancer following treatment with trastuzumab-based therapy. In preclinical models, neratinib has shown evidence of activity against models of NF2-deficient tumors.

  - It is expected that 20 people will take part in the Neratinib Sub-study. A minimum of 2 subjects per tumor type (vestibular schwannoma, non-vestibular schwannoma, meningioma, and ependymoma) must be accrued. Analysis will be performed to determine the radiographic response rate (RR) for each tumor types.
* A subset of 5 participants will be enrolled into the PET imaging biomarker study. These participants will have additional PET scans performed just prior to the first dose of neratinib and after starting the treatment (witin 24 to 72 hours).

ELIGIBILITY:
Eligibility Specific For MASTER PROTOCOL:

Inclusion Criteria:

- Patients must have a pathogenic variant in the NF2 gene (either in the germline or in two NF2-related tumors) OR a confirmed diagnosis of NF2 by fulfilling National Institute of Health (NIH) criteria or Manchester criteria:

The NIH criteria includes presence of:

* Bilateral vestibular schwannomas, OR
* First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity.

The Manchester criteria includes presence of:

* Bilateral vestibular schwannomas, OR
* First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity, OR
* Unilateral vestibular schwannoma AND any two of: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity, OR
* Multiple meningiomas (two or more) AND unilateral vestibular schwannoma OR any two of: schwannoma, glioma, neurofibroma, cataract.

Subjects must have a target NF2-related tumor (VS, non-VS, meningioma, or ependymoma) with documented radiographic progression within the preceding 36 months of Master Study registration defined as either:

* at least 20% increase in volume of enhancing tumor
* at least 2 mm increase in greatest linear dimension of enhancing tumor

Participants must have measurable disease, defined as:

* VS, non-VS, or meningioma target lesions that can be accurately measured as at least 1 ml by volumetric MRI scan or in at least one dimension as ≥10 mm with conventional MRI scan. See protocol for the evaluation of measurable disease
* Ependymoma target lesions measurable linearly.

Participant must have a target NF2-related tumor with the following qualities:

* Not amenable to surgery due to patient refusal or due to high risk for surgical complications (e.g., damage to nerve function). Participant must be ≥ 12 years of age on Day 1 of treatment. Life expectancy of greater than 1 year Karnofsky performance status ≥ 70 or ECOG PS 0 or 1 (see Appendix A). Ability to understand and the willingness to sign written informed consent and assent documents.
* Must have established relationship with primary care physician and provide contact information

Exclusion Criteria:

* Participants who have had chemotherapy within a minimum of 4 weeks prior to Master Study registration (or a minimum of 5 half-lives and resolution to baseline of toxicities unless there are irreversible toxicities from prior drug that do not influence risk of next drug).
* Participants who have received radiation to the target tumor within the last 3 years prior to Master study registration.
* Participants who are receiving any other investigational agents.
* Participants with target or non-target nervous system tumors that, in the opinion of the treating investigator, are likely to require active treatment (including surgery) within 6 months of registration to the Master Study.
* History of a different malignancy, unless (a) have been disease-free for at least 2 years and are deemed by the treating investigator to be at low risk for recurrence of that malignancy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the experimental agents may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these experimental agents, breastfeeding should be discontinued if the mother is treated.

Eligibility Criteria Specific to SUB-STUDY A (Brigatinib arm): CLOSED TO ENROLLMENT

Inclusion criteria

* Participants must meet all eligibility criteria outlined in the Master Study
* Participants must be willing and able to provide written informed consent/assent for the brigatinib arm of the INTUITT-NF2 trial.
* Participant is ≥ 12 years of age and has body weight at least 40 kg on Day 1 of treatment.
* Patient must be able to swallow pills.
* Clinical laboratory values as specified below within 28 days before the first dose of study drug, as described in the protocol document:
* Female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Non-sterilized female patients of reproductive age group and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below:

Female patients must meet 1 of the following:

* Postmenopausal for at least 1 year before the screening visit, or
* Surgically sterile, or
* If they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing of the informed consent form through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse. Brigatinib may decrease effectiveness of hormonal contraceptives, therefore, women are recommended to use non-hormonal methods of contraception. Highly effective non-hormonal birth control for women of child bearing potential with male partners includes:

  * Sexual abstinence (no sexual intercourse)
  * Intrauterine device (IUD) or intrauterine system (IUS)
  * Bilateral tubal ligation (both tubes tied)
  * Vasectomized partner

Male patients, even if surgically sterilized (i.e., status post-vasectomy) must agree to 1 of the following:

- Practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or completely abstain from heterosexual intercourse.

Exclusion criteria:

* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug (if applicable)
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Treatment with any investigational products within 1 month or 5 half-lives (whichever is longer) before the first dose of study drug
* Had major surgery within 30 days of the first dose of brigatinib. Minor surgical procedures such as catheter placement or minimally invasive biopsies are allowed.
* Have significant, uncontrolled, or active cardiovascular disease (as outlined in the protocol):
* Have uncontrolled hypertension (defined as an average systolic blood pressure >160 or an average diastolic blood pressure >100 for adults; for children: please refer to table in protocol

Eligibility Criteria Specific to SUB-STUDY B (Neratinib arm):

* Participants must be willing and able to provide written informed consent/assent for the neratinib arm of the INTUITT-NF2 trial.
* Participant must be ≥ 12 years of age and have body weight ≥ 40 kg on Day 1 of treatment.
* Patient must be able to swallow pills.
* Recovery (ie, to Grade 1 or baseline) from all clinically significant AEs related to prior therapies (excluding alopecia, neuropathy, and nail changes).
* Clinical laboratory values as specified below within 14 days before the first dose of study drug:
* ALT/aspartate aminotransferase (AST) ≤ 2.5 × institutional upper limit of normal (ULN);
* Total serum bilirubin ≤ 1.5 × institutional ULN (<3.0 × institutional ULN for patients with Gilbert syndrome)
* Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2, using the modification of diet in renal disease (MDRD) equation
* Serum lipase ≤1.5 × institutional ULN
* Absolute neutrophil count ≥1.5 × 109/L
* Platelet count ≥75 × 109/L
* Hemoglobin ≥9 g/dL
* Left ventricular ejection fraction (LVEF) ≥50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
* It is not known what effects neratinib has on human pregnancy or development of the embryo or fetus. Therefore, female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Non-sterilized female patients of reproductive age group and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below:

Female patients must meet 1 of the following:

* Postmenopausal for at least 1 year before the screening visit, or
* Surgically sterile, or
* If they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing of the informed consent form through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse. Neratinib may decrease effectiveness of hormonal contraceptives, therefore, women are recommended to use non-hormonal methods of contraception. Highly effective non-hormonal birth control for women of child bearing potential with male partners includes:

  * Sexual abstinence (no sexual intercourse)
  * Intrauterine device (IUD) or intrauterine system (IUS)
  * Bilateral tubal ligation (both tubes tied)
  * Vasectomized partner

Male patients, even if surgically sterilized (i.e., status post-vasectomy) must agree to 1 of the following:

* Practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or completely abstain from heterosexual intercourse.
* Female patients must have negative β-human chorionic gonadotropin (hCG) pregnancy test for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after menopause. [Women are considered postmenopausal if they are ≥12 months without menses, in the absence of endocrine or anti-endocrine therapies.]

Exclusion Criteria

* Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug (if applicable)
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Treatment with any investigational products within 28 days or 5 half-lives (whichever is longer) before the first dose of study drug
* Had major surgery within 30 days of the first dose of neratinib. Minor surgical procedures such as catheter placement or minimally invasive biopsies are allowed.
* Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:
* Myocardial infarction within 6 months before the first dose of neratinib.
* Unstable angina within 6 months before first dose of neratinib.
* Congestive heart failure within 6 months before first dose of neratinib.
* History of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician.
* Any history of clinically significant ventricular arrhythmia.
* Had a cerebrovascular accident or transient ischemic attack within 6 months before first dose of neratinib.
* QTc interval >0.450 seconds (males) or >0.470 (females), or known history of QTc prolongation or Torsade de Pointes (TdP)
* Have a known history of HIV infection. Testing is not required in the absence of history.
* Have malabsorption syndrome or other GI illness that could affect oral absorption of neratinib. Note: This includes any predisposing chronic condition resulting in baseline grade 2 or higher diarrhea
* History of severe allergic reactions or intolerability attributed to compounds of similar chemical or biologic composition to neratinib.
* Have any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of neratinib.
* Concurrent use of enzyme-inducing antiepileptic drugs (EIAEDs), including phenytoin, carbamazepine, oxcarbazepine, fosphenytoin, phenobarbital, pentobarbital, or primidone
* Received systemic treatment with certain cytochrome P-450 inhibitors or inducers within 14 days before enrollment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic response rate (for each drug substudy) | 2 years
  Radiographic response rates in target tumors according to tumor-associated criteria:
  * VS, non-VS, and meningiomas: Dombi criteria (2013)
  * Ependymomas: RECIST 1.12

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability | 2 years
  Number of Participants with Treatment Emergent Adverse Events as Assessed CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Scott Plotkin, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - University of Miami, Miami, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University Langone Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Plotkin SR, Yohay KH, Nghiemphu PL, Dinh CT, Babovic-Vuksanovic D, Merker VL, Bakker A, Fell G, Trippa L, Blakeley JO; INTUITT-NF2 Consortium. Brigatinib in NF2-Related Schwannomatosis with Progressive Tumors. N Engl J Med. 2024 Jun 27;390(24):2284-2294. doi: 10.1056/NEJMoa2400985. Epub 2024 Jun 21. PMID 38904277